CLINICAL TRIAL: NCT00524030
Title: A Double-Blind, Randomized, Multicenter Efficacy And Safety Study Of Pregabalin (Lyrica) As Monotherapy In Patients With Partial Seizures
Brief Title: Efficacy And Safety Study Of Pregabalin (Lyrica) As Monotherapy In Patients With Partial Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081047
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2018-12

CONDITIONS: Epilepsies, Partial
Keywords: Epilepsy; partial seizures; pregabalin monotherapy; double-blind and randomized trial
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: pregabalin 600 mg/day
- 2 (Experimental)
  Interventions: Drug: pregabalin 150 mg/day

INTERVENTIONS:
Drug: pregabalin 600 mg/day — pregabalin 600 mg/day (300mg BID), duration is 20 weeks.
  Arms: 1
Drug: pregabalin 150 mg/day — pregabalin 150 mg/day (75mg BID), duration is 20 weeks.
  Arms: 2

SUMMARY:
This study will determine the safety and efficacy of pregabalin (Lyrica) when administered by itself (without any other anti-epileptic medication) to epilepsy subjects for the treatment of partial seizures. The duration of the trial is about 6 months.

DETAILED DESCRIPTION:
After review of the interim analysis results, the independent Data Monitoring Committee (DMC) recommended to stop the study based on positive efficacy findings for the primary efficacy endpoint according to pre-specified stopping rules. Pfizer accepted the DMC recommendation and made the decision to stop the study on September 7, 2011.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy with partial seizures.
* Males or females, age 18 years or older.
* Documented history of at least 4 partial seizures in the 8 weeks prior to the screening visit.
* Stable treatment with 1 to 2 anti-epileptic drugs in the 8 weeks prior to the screening visit.

Exclusion Criteria:

* Current diagnosis of febrile seizures or seizures related to an ongoing acute medical event.
* Seizures occurring only in cluster patterns, or seizures of a metabolic, toxic or infectious origin.
* Primary generalized epilepsy or status epilepticus within the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2007-09; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (61):
- United States (53):
  - Pfizer Investigational Site, Northport, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Murrieta, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Suwanee, Georgia
  - Pfizer Investigational Site, Anderson, Indiana
  - Pfizer Investigational Site, Danville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Bowling Green, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Houma, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Pikesville, Maryland
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Hattiesburg, Mississippi
  - Pfizer Investigational Site, Great Falls, Montana
  - Pfizer Investigational Site, Cedarhurst, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Rocky Mount, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Indiana, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Czechia (3):
  - Pfizer Investigational Site, Beroun
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Litomyšl
- Pfizer Investigational Site, New Territories, Hong Kong
- Ukraine (4):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Luhansk
  - Pfizer Investigational Site, Odesa

REFERENCES:
- [Derived] French J, Kwan P, Fakhoury T, Pitman V, DuBrava S, Knapp L, Yurkewicz L. Pregabalin monotherapy in patients with partial-onset seizures: a historical-controlled trial. Neurology. 2014 Feb 18;82(7):590-7. doi: 10.1212/WNL.0000000000000119. Epub 2014 Jan 10. PMID 24415567

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin 150 mg/Day: Pregabalin 75 milligram (mg) capsules, administered orally twice daily (BID), for up to a 20-week Double-Blind Treatment Phase, which included an 8-week conversion period (antiepileptic drug [AED] taper) and a 12-week pregabalin Monotherapy Period, followed by a 1-week Titration/Taper phase.
- Pregabalin 600 mg/Day: Pregabalin 300 mg capsules, administered orally, BID for up to a 20-week Double-Blind Treatment Phase, which included an 8-week conversion period (2-week pregabalin dose escalation/6-week AED taper) and a 12-week pregabalin Monotherapy Period, followed by a 1-week Titration/Taper phase. Dose escalation to 600 mg/day occurred over 2 weeks as follows: 75 mg BID on Days 1-7, 150 mg BID on Days 8-14, and 300 mg BID from Day 15 up to Week 20.
Period: Overall Study
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Started | 32 | 129
Completed Double-Blind Treatment Phase | 15 | 70
Completed Taper/Titration Phase | 15 | 70
Completed | 15 | 70
Not Completed | 17 | 59
Not completed — Lack of Efficacy | 10 | 24
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Noncompliance/Investigator discretion | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 3 | 21
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day | Total
Number analyzed (Participants) | 32 | 129 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (12.4) | 39.9 (13.2) | 39.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 71 | 89
  Male | 14 | 58 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the Pregabalin 600 mg/Day Treatment Group Discontinuing the Study Due to at Least 1 Pre-Defined Seizure Exit Criteria
Description: Participants who discontinued due to: episode of status epilepticus (SE); secondarily generalized tonic-clonic (SGTC) seizure if none within 2 years of study entry; 28-day study seizure rate during double-blind phase (DBP) greater than (>)2 times maximum (Max) 28-day study seizure rate during baseline phase (BLP); 2-day study seizure rate during DBP >2 times Max 2-day study seizure rate during BLP; or unacceptable clinically significant increase in frequency/intensity of seizure activity. Determined as exit rate:(1-Kaplan-Meier [KM] product limit estimate for survival function) * 100%
Time Frame: Week 2 up to Week 18
Population: Modified Intent to Treat (MITT) Efficacy Set: The first 125 participants randomized who received at least 1 dose of pregabalin in DB treatment phase, had BL seizure assessment, and participated in DB efficacy assessment after Week 2. Number of participants analyzed (N)= number of MITT participants with discontinuation/completion data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pregabalin 600 mg/Day
Number analyzed (Participants) | 102
Percentage of Participants | 31.9 [20.7 to 43.1]
Statistical Analysis 1: Comparison: Pregabalin 600 mg/Day; Null hypothesis (H0): Exit rate greater than or equal to (≥)74%; Test type: Superiority or Other; p < 0.001, Wald Test; 2-sided 95% adjusted confidence interval constructed using KM product limit estimation and Greenwood's formula for variance with continuity correction
Statistical Analysis 2: Comparison: Pregabalin 600 mg/Day; H0: Exite rate ≥68%; Test type: Superiority or Other; p < 0.001, Wald Test; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants in the Pregabalin 150 mg/Day Treatment Group Discontinuing the Study Due to at Least 1 Pre-Defined Seizure Exit Criteria
Description: Participants who discontinued due to: episode of SE; SGTC seizure if none within 2 years of study entry; 28-day study seizure rate during DBP >2 times Max 28-day study seizure rate during BLP; 2-day study seizure rate during DBP >2 times Max 2-day study seizure rate during BLP; or unacceptable clinically significant increase in frequency/intensity of seizure activity. Determined as exit rate, defined as (1-KM product limit estimate for survival function) * 100%
Time Frame: Week 2 up to Week 18
Population: MITT Full Study Set: all randomized participants who met the MITT definition (received at least 1 dose of pregabalin in DB treatment phase, had BL seizure assessment, and participated in DB efficacy assessment after Week 2)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pregabalin 150 mg/Day
Number analyzed (Participants) | 28
Percentage of Participants | 37.7 [15.4 to 60]
Statistical Analysis 1: Comparison: Pregabalin 150 mg/Day; H0: Exit rate ≥74%; Test type: Superiority or Other; p < 0.001, Wald test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin 150 mg/Day; H0: Exit rate ≥68%; Test type: Superiority or Other; p = 0.001, Wald test; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Completing 20 Weeks of Double-Blind Treatment
Time Frame: Randomization up to Week 20
Population: MITT Full Study Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 28 | 120
Percentage of Participants | 53.6 | 58.3

4. Secondary Outcome: Percentage of Participants Who Met Protocol-Specified Exit Events
Description: Percentage of participants experiencing any of the following (could have had more than 1): 1) episode of SE; 2) SGTC seizure if none had been experienced within 2 years of study entry; 3) 28-day study seizure rate during DBP >2 times the Max 28-day study seizure rate during BLP; 4) 2-day study seizure rate during the DBP >2 times the Max 2-day study seizure rate during BLP; or 5) unacceptable clinically significant increase in frequency/intensity of seizure activity
Time Frame: Week 2 up to Week 18
Population: MITT Efficacy Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 23 | 102
Percentage of Participants
  Status Epilepticus | 0 | 1.0
  SGTC Seizure (not experienced in previous 2 years) | 0 | 2.9
  28-Day Seizure Rate >2 times Max Baseline Rate | 13.0 | 10.8
  2-Day Seizure Rate >2 times Max Baseline Rate | 13.0 | 7.8
  Increased Frequency/Intensity of Seizure Activity | 17.4 | 14.7
  Total | 39.1 | 28.4

5. Secondary Outcome: Mean Time on Pregabalin Monotherapy
Time Frame: Week 2 to Week 20
Population: MITT Full Study Set; N=number of participants entering Monotherapy Period
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 22 | 97
Days | 73.8 (30.15) | 78.0 (28.24)

6. Secondary Outcome: Percentage of Seizure-Free Participants by Study Phase
Description: Percentage of participants who were seizure-free during the last 28 days on double-blind study medication (monotherapy phase, Days 112-140), during the monotherapy portion of the double-blind treatment phase (Days 56-140), and during all of the double-blind treatment phase (Days 1-140)
Time Frame: Day 1 up to Day 140
Population: MITT Full Study Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 28 | 120
Percentage of Participants
  Last 28 Days of Monotherapy (Days 112-140) | 17.9 | 12.5
  Monotherapy (Days 56-140) | 7.1 | 6.7
  Entire Double-Blind Treatment (Days 1-140) | 0 | 1.7

7. Secondary Outcome: Pregabalin Population Pharmacokinetics (PK)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Baseline up to 20 weeks
Population: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pregabalin Exposure-Response Analysis
Description: Percentage of participants predicted to exit the study due to any seizure exit criteria at Day 126. The exit rate at Day 126 was predicted using the final model (log normal distribution with respect to treatment group) and the parameter estimates.
Time Frame: Day 126
Population: MITT Full Study Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Number analyzed (Participants) | 28 | 120
Percentage of Participants | 37.2 | 26.3

ADVERSE EVENTS:
Time Frame: Baseline to Week 21
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 600 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/32 | 17/129
Other Adverse Events (participants affected / at risk) | 15/32 | 75/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 150 mg/Day (N=32) | Pregabalin 600 mg/Day (N=129)
Angina pectoris (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Complex partial seizures (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 5
Epilepsy (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 150 mg/Day (N=32) | Pregabalin 600 mg/Day (N=129)
Vision blurred (Eye disorders) | 1 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 8
Fatigue (General disorders) | 2 | 20
Oedema peripheral (General disorders) | 1 | 8
Alanine aminotransferase increased (Investigations) | 2 | 1
Weight increased (Investigations) | 2 | 21
Balance disorder (Nervous system disorders) | 0 | 8
Disturbance in attention (Nervous system disorders) | 3 | 4
Dizziness (Nervous system disorders) | 5 | 25
Dysarthria (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 0 | 13
Somnolence (Nervous system disorders) | 5 | 22
Confusional state (Psychiatric disorders) | 0 | 7

LIMITATIONS AND CAVEATS:
External Data Monitoring Committee (DMC) determined study met criteria to stop early for positive efficacy. Exit rate was the basis for primary analysis and is what is reported here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.